CLINICAL TRIAL: NCT01758653
Title: Carbon Monoxide Blood and DNA Repository
Brief Title: Carbon Monoxide Blood and DNA Biorepository
Status: Enrolling by invitation | Type: Observational
Sponsor: Intermountain Health Care, Inc. (Other)
Responsible Party: Principal Investigator, Lindell Weaver, Lindell Weaver, MD, Intermountain Health Care, Inc.
Other Study IDs: 1024109
Record Dates: First submitted 2012-12-27; First posted 2013-01-01 (Estimated); Last update posted 2023-09-29 (Actual); Status verified 2023-09

CONDITIONS: Carbon Monoxide Poisoning
Keywords: CO poisoning
MeSH Terms: conditions — Carbon Monoxide Poisoning

STUDY DESIGN:
Observational Model: Cohort | Time Perspective: Prospective
Biospecimen Retention: Samples With DNA — Blood for plasma, serum, and DNA sequestration
Oversight: Data Monitoring Committee: No

GROUPS / COHORTS (1):
- Biorepository: Patients with acute CO poisoning. Blood collection for biorepository only, no study intervention.
  Interventions: Other: No study intervention

INTERVENTIONS:
Other: No study intervention — There is no study-related intervention.

SUMMARY:
The purpose of this biorepository is to collect blood from patients at the time of CO poisoning and at follow-up visits months to years later. These samples can be used in the future to learn more about how CO damages the heart and brain and whether blood tests could predict which patients will have problems after CO poisoning.

DETAILED DESCRIPTION:
The investigators propose to establish a biorepository for storage of serum, plasma, and DNA collected from patients with carbon monoxide (CO) poisoning. Participants will also be evaluated for clinical outcome. The biorepository will include serum and plasma from CO-poisoned patients drawn at the time of injury as well as from blood drawn at clinical follow-up visits. The biorepository will also bank DNA from these participants.

These specimens can be analyzed in the future to elucidate potential inflammatory and immunological mechanisms that cause brain and heart damage and identify possible biological and genetic predictors of poor outcome.

ELIGIBILITY:
Inclusion Criteria:

1. Symptomatic carbon monoxide poisoning (headache, nausea, vomiting, dizziness, fatigue, muscle aches, slowed mentation, confusion, loss of consciousness, etc.).
2. Documented exposure to carbon monoxide and no other reasonable explanation for their signs and symptoms.

Exclusion criteria:

1. Pregnancy
2. Age < 18 years
3. Unable to obtain informed consent
4. Subjects who, in the opinion of the investigator, are unable to comply with the requirements of the study or are unsuitable for any reason. The investigator and the Sponsor, prior to enrolling the subject on a case-by-case basis, must approve and document any waiver of these inclusion and exclusion criteria.
5. Anemia requiring blood products within the last 4 months or hematocrit less than the laboratory normal reference range

Min Age: 18 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Study Population: Study population includes patients who present to LDS Hospital or Intermountain Medical Center with symptomatic carbon monoxide poisoning and documented exposure to carbon monoxide.
Sampling Method: Non-Probability Sample
Enrollment: 300 (Estimated)
Dates: Start 2012-02 (Actual); Primary Completion 2032-12 (Estimated); Study Completion 2032-12 (Estimated)

PRIMARY OUTCOMES:
Biorepository for serum and plasma | Within 24 hours of CO Poisoning
  Serum and plasma from blood collected within 24 hours of acute CO poisoning

SECONDARY OUTCOMES:
Serum and plasma (sub-acute) | 4 weeks to 4 months after CO poisoning
  Serum and plasma collected 4 weeks to 4 months after poisoning
DNA Sequestration | 24 hours to 12 months after CO poisoning
  DNA sequestered from blood drawn up to 1 year from CO poisoning
Serum and plasma (long-term) | 4 months to 12 months after CO poisoning
  Serum and plasma collected 4 months to 12 months after poisoning

CONTACTS AND LOCATIONS:
Overall Officials: Lindell K. Weaver, MD, Principal Investigator — Intermountain Health Care, Inc.
Locations (2):
- United States (2):
  - Intermountain Medical Center, Murray, Utah
  - LDS Hospital, Salt Lake City, Utah